CLINICAL TRIAL: NCT02251483
Title: Use of Serum-derived Immunoglobulin/Protein Isolate (SBI) for the Maintenance of Health in Subjects With Irritable Bowel Syndrome (IBS) Following Successful Treatment of Small Intestinal Bacterial Overgrowth (SIBO)
Brief Title: Use of SBI in IBS Subjects Following a Successful Treatment of Small Intestinal Bacterial Overgrowth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Entera Health, Inc (Industry)
Responsible Party: Principal Investigator, Mark Pimentel, MD, Director, GI Motility Program, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 35543
Record Dates: First submitted 2014-09-17; First posted 2014-09-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Diarrhea Predominant Irritable Bowel Syndrome; Small Intestinal Bacterial Overgrowth
Keywords: DIBS; SIBO

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SBI (Other): Group 1: SBI (N=30) - one packet daily
  Interventions: Other: Serum-derived bovine immunoglobulin protein isolate (SBI)
- Placebo (Placebo Comparator): Group 2: Placebo (N=30) - one packet daily
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Serum-derived bovine immunoglobulin protein isolate (SBI)
  Arms: SBI
Other: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine whether giving SBI as a medical food starting with maintenance of health in the management of chronic loose and frequent stools in IBS-D subjects with SIBO after successful treatment with rifaximin can lead to more prolonged duration of benefit and delay symptom recurrence. SBI is the main ingredient in EnteraGam™, an orally administered prescription medical food for the dietary management of patients with enteropathy or chronic loose or frequent stools, including patients with IBS-D.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is one of the most common gastrointestinal disorders, with a global prevalence of 11%. IBS manifests itself in 3 major forms; diarrhea-predominant (IBS-D), constipation-predominant (IBS-C), and mixed (IBS-M), and is predominantly characterized by symptoms of abdominal pain, changes in stool frequency and consistency, and abdominal bloating.

SIBO is a condition in which there is an increase in the number of bacteria in the small bowel, and typically includes an overgrowth of coliform bacteria which are normally found in the colon. These ferment carbohydrates into gas (which can be measured using the lactulose breath test (LBT)), and the SIBO hypothesis proposes that it is this expansion of bacteria in the small bowel that leads to IBS symptoms including bloating, abdominal discomfort and changes in stool form. The antibiotic rifaximin is used to treat IBS-D, and has been shown to normalize the LBT in 70% of subjects. Despite this success, symptoms such as SIBO tend to recur, usually within 4 months of finishing the antibiotic treatment. Therefore, there remains a significant need to identify therapeutic agents which can maintain the health of subjects with IBS and SIBO and increase the duration of benefit in subjects with IBS and SIBO following antibiotic treatment.

SBI is intended for the dietary management of enteropathy under medical supervision in patients with chronic loose or frequent stools, including IBS-D patients. In vitro and animal studies have shown that SBI supports digestive and absorptive properties of the intestinal tracts by:

1. Binding and neutralizing microbial components
2. Helping to maintain beneficial gut microbiota
3. Managing gut barrier function
4. Maintaining GI immune balance

Clinical studies have also demonstrated that oral SBI improves nutrient absorption, nutritional status and GI symptoms in patients with HIV-associated enteropathy, IBS-D, or malnutrition. It is important to note that SBI is not used to treat patients with IBS-D or other enteropathies, but is given as a medical food to assist in the maintenance of health only.

This study will assess whether giving SBI as a medical food to subjects with IBS-D and SIBO after they successfully complete a course of rifaximin can lead to more prolonged maintenance of health and duration of benefit of antibiotic treatment in IBS-D patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-75 years old
* Meet Rome II criteria for IBS-D
* Meet criteria for SIBO
* If ≥50 years old, a colonoscopy must have been completed within the past 10 years
* Have just completed a course of antibiotic treatment with rifaximin and successfully responded to this treatment.

Exclusion Criteria:

* Had intestinal surgery (except appendectomy or cholecystectomy)
* Pelvic floor dysfunction
* Pregnancy or nursing mothers
* History of bowel obstruction
* History of celiac disease
* History of inflammatory bowel disease
* Cirrhosis
* Diabetes
* Use of tricyclic antidepressants
* Use of antidiarrheal medications
* Allergy or hypersensitivity to beef or any component of SBI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Time to relapse (symptom recurrence) in subjects with IBS-D after successful treatment with rifaximin | up to 4 months

SECONDARY OUTCOMES:
Change in symptoms based on comparison of baseline symptom questionnaire to weekly symptom questionnaires | baseline and weekly questionnaires for up to 4 months
Comparison of baseline Bristol stool score based on 7 day stool diary | last week of every month for up to 4 months
Comparison of KT ratios in plasma samples | up to 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- GI Motility Program Cedars-Sinai Medical Center, Los Angeles, California, United States